CLINICAL TRIAL: NCT00211185
Title: A Pilot Phase II Study to Determine the Safety and Efficacy of the Combination of ONTAK With CHOP in Peripheral T-Cell Lymphoma.
Brief Title: A Study of ONTAK and CHOP in Newly Diagnosed, Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #35
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — denileukin diftitox; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; pegfilgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denileukin diftitox in combination with CHOP (Experimental): Unblinded denileukin diftitox at 18 micrograms/kilogram/day (ug/kg/d) was administered intravenously (IV) on Days 1 and 2 of each 21-day cycle. Cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) was administered on Day 3 of each 21-day cycle. On Day 4 of each 21-day cycle, pegfilgrastim (a granulocyte colony-stimulating factor (G-CSF)) was started as a prophylaxis to prevent neutropenia. After completion of two 21-day cycles, participants were evaluated for clinical response. Two 21-day cycles with denileukin and CHOP were repeated followed by response evaluations after each set of two 21-day cycles with intent to treat for 6 cycles, with a maximum of 8 cycles.
  Interventions: Drug: Denileukin diftitox; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Other: Pegfilgrastim

INTERVENTIONS:
Drug: Denileukin diftitox — Denileukin diftitox will be administered intravenously (IV) at a dosage of 18 micrograms/kilogram/day (ug/kg/d) on Days 1 and 2 of each 21-Day cycle for a total of 6 cycles, with a maximum of 8 cycles.
  Other Names: ONTAK; DAB389 IL-2
Drug: Cyclophosphamide — Cyclophosphamide will be administered IV at a dosage of 750 milligrams/meter squared (mg/m^2) on Day 3 of each 21-day cycle for 6 cycles, with a maximum of 8 cycles.
  Other Names: CHOP
Drug: Doxorubicin — Doxorubicin will be administered IV at a dosage of 50 mg/m^2 on Day 3 of each 21-day cycle for 6 cycles, with a maximum of 8 cycles.
  Other Names: CHOP
Drug: Vincristine — Vincristine will be administered IV at a dosage of 1.4 mg/m^2 on Day 3 of each 21-day cycle for 6 cycles, with a maximum of 8 cycles.
  Other Names: CHOP
Drug: Prednisone — Prednisone will be administered orally at a dosage of 100 mg on Days 3 to 7 of each 21-day cycle for 6 cycles, with a maximum of 8 cycles.
  Other Names: CHOP
Other: Pegfilgrastim — Pegfilgrastim will be administered at a dosage of 6 mg subcutaneously on Day 4 to help prevent neutropenia. Alternatively, participants received filgrastim 5 ug/kg/d starting on Day 4 and continued until absolute neutrophil count (ANC) was less than 5000/millimeter squared (mm^2) for 2 days post-nadir.
  Other Names: Neulasta; granulocyte-colony stimulating factor; G-CSF

SUMMARY:
Study of ONTAK and CHOP (chemotherapy drugs) to find out their ability to make Peripheral T-cell lymphoma disappear (for any period of time) and potentially lengthen life. The study will also compare what kind of side effects these drugs cause and how often they occur. The hypothesis is that patients with newly diagnosed peripheral T-Cell lymphoma, when given ONTAK + CHOP, will tolerate the treatment and will have a 20% improvement in response rate when compared to CHOP alone.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of peripheral T-cell lymphoma of one of the following histologies as per the REAL classification: peripheral T-cell lymphoma (unspecified), anaplastic large cell lymphoma CD30+, angioimmunoblastic T-cell lymphoma, nasal/nasal type T/NK cell lymphoma, intestinal T-cell lymphoma, hepatosplenic T-cell lymphoma, subcutaneous panniculitic T-cell lymphoma.
* Treatment naïve except for prior radiation or a single cycle of CHOP.
* Patients must have at least one clear-cut bidimensionally measurable site by physical exam and/or computed tomography.
* Prior radiation therapy for localized disease is allowed as long as the irradiated area is not at the mediastinal area or at the only site of measurable disease. Therapy must be completed at least 4 weeks before the enrollment in study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* At least 18 years of age.
* Adequate bone marrow reserve, indicated by absolute neutrophil count (ANC) > or equal to 1000/microL, platelets > or equal to 50,000/microL (25,000/MicroL if thrombocytopenia secondary to bone marrow involvement by lymphoma), and hemoglobin > or equal to 8 g/dL.
* Adequate liver function, indicated by bilirubin < or equal to 1.5 times the upper limit of normal (ULN), alanine transaminase (ALT) < or equal to 2 times the ULN or aspartate transaminase (AST) < or equal to 2.0 times the ULN, and albumin > or equal to 3.0 g/dL.
* Adequate renal function, indicated by serum creatinine < or equal to 2.5 mg/dL.
* Women of childbearing potential and sexually active males agree to use an accepted and effective method of contraception.
* Able to give informed consent.

Exclusion Criteria:

* Diagnosis of Mycosis Fungoides or Sezary Syndrome.
* Active Hepatitis B or Hepatitis C infection.
* Known HIV infection (HIV testing is not required).
* Patients with active infections requiring specific anti-infective therapy are not eligible until all signs of infections have resolved and any continuing treatment if appropriate is given on an outpatient basis.
* Previous doxorubicin therapy with cumulative dose of >100 mg/m2.
* Left Ventricular Ejection Fraction (LVEF) < 50%.
* Patients who are pregnant or breast-feeding.
* Prior invasive malignancies within past 5 years.
* Allergy to or history of allergy to diphtheria toxin or IL-2.
* Preexisting severe cardiovascular disease (e.g. CHF, Severe CAD, cardiomyopathy, MI within the past 3 months, arrhythmia) requiring ongoing treatment.
* Ongoing antineoplastic chemotherapy, radiation, hormonal (excluding contraceptives) or immunotherapy, or investigational medications within past 30 days.
* Patients with deep vein thrombosis within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-03-14 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2009-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Siouxland Hematology Oncology, Sioux City, Iowa
  - Kansas City Cancer Centers, Lenexa, Kansas
  - Dana Farber/ Harvard Cancer Center, Boston, Massachusetts
  - New England Medical Center, Boston, Massachusetts
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Kansas City Cancer Centers, Kansas City, Missouri
  - St. Joseph Oncology Inc., Saint Joseph, Missouri
  - Arch Medical Services, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology Oncology Associates of NNJ, Morristown, New Jersey
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Barrett Cancer Center-University of Cincinnati, Cincinnati, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Cancer Center, Arlington, Texas
  - Marnie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology,P.A., Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - The Texas Cancer Center, Dallas, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, Garland, Texas
  - Longview Cancer Center, Longview, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - HOAST Medical Dr., San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer Care and Research Center, Waco, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology and Hematology Associates of SW VA Inc., Salem, Virginia
  - Puget Sound Cancer Center, Edmonds, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- [Result] Francine M. Foss, Nelida Sjak-Shie, Andre Goy, Ranjana Advani, Eric Jacobsen, and Mark Acosta A Phase II Study of Denileukin Diftitox (Ontak®) with CHOP Chemotherapy in Patients with Newly-Diagnosed Aggressive T-Cell Lymphomas, the CONCEPT Trial: Interim Analysis. Blood (ASH Annual Meeting Abstracts), Nov 2006; 108: 2461.
- [Derived] Foss FM, Sjak-Shie N, Goy A, Jacobsen E, Advani R, Smith MR, Komrokji R, Pendergrass K, Bolejack V. A multicenter phase II trial to determine the safety and efficacy of combination therapy with denileukin diftitox and cyclophosphamide, doxorubicin, vincristine and prednisone in untreated peripheral T-cell lymphoma: the CONCEPT study. Leuk Lymphoma. 2013 Jul;54(7):1373-9. doi: 10.3109/10428194.2012.742521. Epub 2013 Jan 29. PMID 23278639

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denileukin Diftitox in Combination With CHOP
Started | 49
Completed | 29
Not Completed | 20
Not completed — Death | 2
Not completed — Disease progression | 7
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all treated participants. Participants who did not receive at least 1 dose of study treatment were excluded from this population.
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Summary of All Adverse Events by Frequency in Greater Than 20% of Treated Participants
Description: An adverse event (AE) was any medical occurrence in a participant who was administered denileukin diftitox and cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP), and did not necessarily have a causal relationship with this treatment. An AE included any side effect, injury, toxicity, sensitivity reaction, or any undesirable clinical or laboratory event that was not normally observed in the participant. Safety was assessed for all participants who received at least one dose of study medication and was monitored throughout the study. Safety evaluations were based on the incidence, intensity, and type of AE, and clinically significant changes in the participant's medical history, physical examination findings, vital signs, and clinical laboratory results. Participants also notified the study staff of any problems that occurred between visits by telephone, and if necessary, were evaluated by the investigator or study staff at an unscheduled interim visit.
Time Frame: From date of first dose up to approximately 4 weeks after discontinuation of denileukin diftitox and CHOP, or after early withdrawal for any reason, up to approximately 5 years 9 months
Population: The Safety Population was used and defined as all treated participants. Participants who did not receive at least one dose of study medication were excluded from this population. For this study, the safety population is the same as the Intent to Treat (ITT) population.
Measure: Number; unit: Percentage of participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Percentage of participants
  Fatigue | 63.3
  Nausea | 46.9
  Hemoglobin | 40.8
  Neuropathy-sensory | 40.8
  Alanine transaminase | 34.7
  Hyperglycemia | 34.7
  Hypoalbuminemia | 34.7
  Leukocytes | 34.7
  Fever | 32.7
  Hypocalcemia | 30.6
  Lymphopenia | 30.6
  Aspartate transaminase | 28.6
  Dyspnea | 28.6
  Platelets | 28.6
  Alopecia | 26.5
  Neutrophils | 26.5
  Constipation | 24.5
  Edema-limb | 20.4
  Hyponatremia | 20.4

2. Primary Outcome: Summary of All Treatment-Related Adverse Events by Frequency in Greater Than 10% of Treated Participants
Description: A treatment-related adverse event was any medical occurrence in a participant who was administered denileukin diftitox and CHOP and was determined to be possibly, probably, or definitely related to study treatment. An AE included any side effect, injury, toxicity, sensitivity reaction, or any undesirable clinical or laboratory event that was not normally observed in the participant. Safety was assessed for all participants who received at least one dose of study medication and was monitored throughout the study. Safety evaluations were based on the incidence, intensity, and type of AE, and clinically significant changes in the participant's medical history, physical examination findings, vital signs, and clinical laboratory results. Participants also notified the study staff of any problems that occurred between visits by telephone, and if necessary, were evaluated by the investigator or study staff at an unscheduled interim visit.
Time Frame: as for outcome 1
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Percentage of participants
  Fatigue | 55.1
  Nausea | 36.7
  Hemoglobin | 30.6
  Leukocytes | 30.6
  Lymphopenia | 30.6
  Dyspnea | 26.5
  Neuropathy-sensory | 26.5
  Alanine transaminase | 24.5
  Alopecia | 22.4
  Platelets | 22.4
  Neutrophils | 20.4
  Constipation | 18.4
  Hypoalbuminemia | 18.4
  Aspartate transaminase | 16.3
  Edema-limb | 16.3
  Fever | 16.3
  Hypocalcemia | 16.3
  Allergic reaction | 12.2
  Anorexia | 12.2
  Taste alteration | 12.2
  Febrile neutropenia | 10.2

3. Primary Outcome: Summary of Treatment-Related Adverse Events Greater Than or Equal to Grade 3 by System Organ Class
Description: Treatment-related AEs were medical occurrences determined to be possibly, probably, or definitely related to study treatment. Severity grading of the AE was according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) severity scale (grades 1 - 5) with grade 3 representing a severe AE. Safety was assessed for all participants who received at least one dose of study medication and was monitored throughout the study. Safety evaluations were based on the incidence, intensity, and type of AE, and clinically significant changes in the participant's medical history, physical examination findings, vital signs, and clinical laboratory results. Participants also notified the study staff of any problems that occurred between visits by telephone, and if necessary, were evaluated by the investigator or study staff at an unscheduled interim visit.
Time Frame: as for outcome 1
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Percentage of participants
  Allergy/Immunology: Allergic reaction | 2.0
  Blood/Bone Marrow: Hemoglobin | 8.2
  Blood/Bone Marrow: Leukocytes | 16.3
  Blood/Bone Marrow: Lymphopenia | 24.5
  Blood/Bone Marrow: Neutrophils | 16.3
  Blood/Bone Marrow: Platelets | 12.2
  Cardiac Arrhythmia: Supra Arrhyth:Sinus Tachy | 2.0
  Cardiac General: Cardiac ischemia/infarction | 2.0
  Cardiac General: Cardiopulmonary arrest | 2.0
  Coagulation: Coagulation-other | 2.0
  Constitutional symptoms: Fatigue | 2.0
  Constitutional symptoms: Fever | 2.0
  Death: Death, NOS | 2.0
  Infection: Febrile neutropenia | 10.2
  Infection: Inf, 3-4 ANC: cath-related | 2.0
  Infection: Infection-other | 2.0
  Infection: Lung Inf, 0-2 ANC: lung | 2.0
  Metabolic/Laboratory: Alanine transaminase (ALT) | 4.1
  Metabolic/Laboratory: Aspartate transaminase (AST) | 4.1
  Metabolic/Laboratory: CPK | 2.0
  Metabolic/Laboratory: Cholesterol | 2.0
  Metabolic/Laboratory: GGT | 2.0
  Metabolic/Laboratory: Hypoalbuminemia | 4.1
  Metabolic/Laboratory: Hypokalemia | 2.0
  Pain: Pain-other | 2.0
  Pulmonary/Upper Respiratory: Dyspnea | 4.1
  Pulmonary/Upper Respiratory: Hypoxia | 2.0
  Pulmonary/Upper Respiratory: Pneumonitis | 2.0
  Syndromes: Tumor Lysis syndrome | 2.0
  Vascular: Thrombosis/embolism | 4.1

4. Primary Outcome: Summary of Study Drug-Related (Possible, Probable, or Definite) Serious Adverse Events
Description: A serious adverse event (SAE) was any AE that occurred at any dose and resulted in any of the following outcomes: death, a life-threatening adverse drug experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that did not result in death, were life-threatening, or required hospitalization were considered a SAE when based upon appropriate medical judgment, jeopardized the participant and required medical or surgical intervention to prevent one of the outcomes listed above. Possibly Related (Poss Rel) applied to AEs judged to be perhaps related to study medication, Probably Related (Prob Rel) applied to AEs judged to have a high degree of certainty as related to study medication, and Definitely Related (Def Rel) related applied to AEs that were judged to be without a doubt related to study medication.
Time Frame: as for outcome 1
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Participants
  Febrile neutropenia (grade 3) Prob Rel | 1
  Febrile neutropenia (grade 3) Poss Rel | 4
  Fever (grade 3) Poss Rel | 1
  Fever (grade 2) Poss Rel | 1
  Thrombosis/embolism (grade 3) Poss Rel | 1
  Neutrophils (grade 3) Poss Rel | 1
  Neutrophils (grade 4) Poss Rel | 3
  Left vent. diastolic dysfunct. (grade 1) Poss Rel | 1
  Allergic reaction (grade 4) Def Rel | 1
  Platelets (grade 4) Prob Rel | 1
  Platelets (grade 4) Poss Rel | 2
  Dyspnea (grade 3) Prob Rel | 1
  Pneumonitis (grade 3) Prob Rel | 1
  Lung Inf, 0-2 ANC: lung (grade 3) Poss Rel | 1
  Leukocytes (grade 4) Poss Rel | 2
  Leukocytes (grade 4) Prob Rel | 1
  Lymphopenia (grade 4) Poss Rel | 2
  Inf, 3-4 ANC: cath-related (grade 3) Poss Rel | 1
  Allergy-other (grade 1) Def Rel | 1
  Infection-other (grade 3) Poss Rrel | 1
  Cardiac ischemia (grade 5) Def Rel | 1
  Tumor lysis syndrome (grade 5) Poss Rel | 1
  Cardiopulmonary arrest (grade 4) Poss Rel | 1
  Supra Arrhyth: Sinus Tachy. (grade 4) Poss Rel | 1
  Death, NOS (grade 5) Poss Rel | 1
  Edema-limb (grade 1) Poss Rel | 1
  Pain-other (grade 3) Poss Rel | 1

5. Secondary Outcome: Overall Response in the Intent To Treat (ITT) Population
Description: Response rate was defined as the percentage of the ITT population who achieved a Complete Response (CR), Unconfirmed Complete Response (CRu), or Partial Response (PR). The International Working Group recommendations on non-Hodgkin's lymphoma response criteria were used to determine response to therapy. Largely, the protocol defined the response criteria as: 1) CR, loss of all detectable clinical and radiographic evidence of disease and disease-related symptoms if present before therapy; 2) CRu, CR with the caveats, response to therapy was accompanied with a 75% reduction in measurable lesion size and/or an indeterminate bone marrow biopsy (if initially positive); and 3) PR, less than or equal to 50% decrease in the sum of the measurements of tumor diameters, no increase in the size of other nodes, liver, or spleen, hepatic or spleen nodules regressed by at least 50%, and/or no new sites of disease.
Time Frame: From the start of the treatment to the date of participant's death assessed up to 5 years 9 months
Population: Intent to treat (ITT) population included all participants who signed an informed consent and were deemed eligible to participate by the investigator based on the screening assessments, and started at least 1 cycle of study treatment. It is the same as the Safety Population (SP) for this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Percentage of participants
  Confirmed complete response | 51.0
  Unconfirmed complete response | 4.1
  Partial response | 10.2
  Stable disease | 6.1
  Disease progression | 4.1
  Early death | 4.1
  Inadequate assessment | 20.4

6. Secondary Outcome: Overall Response in the Efficacy Analyzable (EA) Population
Description: Response rate was defined as the percentage of the EA population who achieved a CR, CRu, or PR. The International Working Group recommendations on non-Hodgkin's lymphoma response criteria were used to determine response to therapy. Largely, the protocol defined the response criteria as: 1) CR, loss of all detectable clinical and radiographic evidence of disease and disease-related symptoms if present before therapy; 2) CRu, CR with the caveats, response to therapy was accompanied with a 75% reduction in measurable lesion size and/or an indeterminate bone marrow biopsy (if initially positive); and 3) PR, less than or equal to 50% decrease in the sum of the measurements of tumor diameters, no increase in the size of other nodes, liver, or spleen, hepatic or spleen nodules regressed by at least 50%, and/or no new sites of disease.
Time Frame: From the start of the treatment to the date of the participant's death assessed up to 5 years 9 months
Population: EA population includes all participants who received at least 2 cycles of study drug treatment, were eligible to participate or ineligible with an exception granted by the principal investigator (PI), had bidimensional lesions at baseline, and had at least 1 disease response assessment form submitted following cycle 2.
Measure: Number; unit: Percentage of participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 37
Percentage of participants
  Confirmed complete response | 67.6
  Unconfirmed complete response | 5.4
  Partial response | 13.5
  Stable disease | 8.1
  Disease progression | 5.4
  Early death | 0.0
  Inadequate assessment | 0.0

7. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the length of time from the first date at which the response criteria were met (taking the earliest date at which a PR, CRu, or the confirmed CR occurred) until the date that recurrent or PD or death was accurately documented, per the criteria defined for progression-free survival (PFS). All participants within the EA population who achieved a response per the criteria defined were included in the duration of the response analysis. Participants lost to follow-up prior to PD or death were censored at the date they were last known to still be responding to treatment. Duration of response was estimated using the Kaplan-Meier method with the median duration of response summarized.
Time Frame: From the date of the first documented CR (confirmed or unconfirmed) or PR until the date of first documentation of recurrent or PD or death, assessed up to 5 years 9 months
Population: EA population
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 32
Months | 29.7 (NA) — 90% confidence interval could not be calculated because high number of participants were censored from the analysis.

8. Secondary Outcome: Progression-Free Survival
Description: PFS was defined as the period of time from treatment start to the first documentation of PD, recurrence, or death. PD was defined as a greater than or equal to 50% increase from baseline in the sum of the products of the greatest diameters of any previously identified abnormal node for PRs or non-responders, or the appearance of any new lesions during or at the end of therapy. PFS was censored at the last date for which the response assessment resulted in the absence of PD for participants who did not demonstrate objective progression or recurrence. Participants who withdrew prior to evidence of disease progression or recurrence, PFS was censored at the last date assessment showed an absence of PD.
Time Frame: From the date of first dose of study drug until date of first documentation of PD, recurrence, or death from any cause, assessed up to 5 years 9 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Weeks | 12.4 (6.1)

9. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall Survival (OS) was defined as the time from the date of registration to the date of the participant's death. OS was determined by reviewing all participant's records every 6 months until the study was administratively closed or all participants died, whichever occurred first. Participants who were lost to follow-up but were still alive at the date of last contact were censored at the date of last contact. Participants who did not have a recorded date of death were censored for OS at the last date at which they were known to be alive.
Time Frame: From date of randomization until death, or administrative close of study, whichever came first, assessed up to 5 years 9 months
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Denileukin Diftitox in Combination With CHOP
Number analyzed (Participants) | 49
Percentage of participants | 63.3

ADVERSE EVENTS:
Time Frame: From date of administration of first dose up to 30 days after the last dose, or for any event that was present prior to study drug and continued after the first dose of study treatment but worsened in intensity, up to approximately 5 years 9 months
Description: Treatment-emergent adverse events and serious adverse events were reported. Safety population included all treated participants. Participants who did not receive at least 1 dose of study treatment were excluded from this population. All toxicities were graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 3.0.
Arm/Group | Denileukin Diftitox in Combination With CHOP
All-Cause Mortality (participants affected / at risk) | 18/49
Serious Adverse Events (participants affected / at risk) | 25/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denileukin Diftitox in Combination With CHOP (N=49)
Allergic reaction (Immune system disorders) | 1
Allergy-other (Immune system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutrophils (Blood and lymphatic system disorders) | 4
Platelets (Blood and lymphatic system disorders) | 3
Supra Arrhyth: Sinus Tachy (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 2
Cardiopulmonary arrest (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Left vent. diastolic dysfunct. (Cardiac disorders) | 1
Fever (General disorders) | 6
Death NOS (General disorders) | 1
Disease progression, NOS (General disorders) | 2
GI obstruction, small bowel (Gastrointestinal disorders) | 1
Lung hemorrhage, lung (General disorders) | 1
Febrile Neutropenia (Infections and infestations) | 6
Inf. 0-2 ANC: cath-related (Infections and infestations) | 1
Inf, 3-4 ANC: blood (Infections and infestations) | 1
Inf, 3-4 ANC: cath-related (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Lung inf, 0-2 ANC: lung (Infections and infestations) | 1
Skin Inf, 0-2 ANC: skin (Infections and infestations) | 1
Edema-limb (General disorders) | 1
Alanine transaminase (AST) (Investigations) | 1
Creatinine phosphokinase (CPK) (Investigations) | 1
Cerebral spinal fluid (CSF) leak (Investigations) | 1
Neurop. lat dev. of eye (Eye disorders) | 1
Cardio. pain cardiac/heart (General disorders) | 1
GI pain, abdomen (General disorders) | 1
Pain-other (General disorders) | 1
Pain NOS (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Tumor lysis syndrome (General disorders) | 1
Thrombosis/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denileukin Diftitox in Combination With CHOP (N=49)
Edema-limb (Blood and lymphatic system disorders) | 9
ALT (Investigations) | 17
Fatigue (General disorders) | 31
Weight gain (General disorders) | 5
Hypocalcemia (Investigations) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 3
Fever (General disorders) | 11
Hypoalbuminemia (Investigations) | 17
Ulceration (Skin and subcutaneous tissue disorders) | 2
AST (Investigations) | 14
Rigors/chills (General disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 15
Constipation (Gastrointestinal disorders) | 12
Hemoglobin (Investigations) | 20
Nausea (Gastrointestinal disorders) | 23
Leukocytes (Investigations) | 17
Neutrophils (Investigations) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 7
Musculoskeletal-other (Musculoskeletal and connective tissue disorders) | 2
Neuropathy-motor (Nervous system disorders) | 3
Incontinence, urinary (Renal and urinary disorders) | 1
Neuro Inf, 0-2 ANC: periph nrv (Infections and infestations) | 2
Alopecia (General disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 6
Alkaline phosphatase (Investigations) | 4
Sweating (General disorders) | 6
Weight loss (General disorders) | 5
Mucositis, funct: oral cav (Infections and infestations) | 2
Proteinuria (Investigations) | 2
Hypokalemia (Investigations) | 6
Muscle weakness: up. extrem. (Musculoskeletal and connective tissue disorders) | 2
Musculo. pain: bone (Musculoskeletal and connective tissue disorders) | 8
Platelets (Investigations) | 14
Hyperglycemia (Investigations) | 16
Hemoglobinuria (Investigations) | 1
Nail changes (General disorders) | 2
Libido (Reproductive system and breast disorders) | 2
Taste alteration (General disorders) | 9
Neuro Pain: head/headache (Nervous system disorders) | 7
Vaginitis (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Thrombosis/embolism (Vascular disorders) | 4
Allergic reaction (Immune system disorders) | 6
Palpitations (Cardiac disorders) | 3
Heartburn (Gastrointestinal disorders) | 8
Hot flashes (General disorders) | 4
Blurred vision (Eye disorders) | 5
Flatulence (Gastrointestinal disorders) | 2
Confusion (Psychiatric disorders) | 2
Cardio. Pain: cardiac/heart (Cardiac disorders) | 2
Left vent. diastolic function (Cardiac disorders) | 1
Mood alterations: depression (Psychiatric disorders) | 4
Skin Inf., 0-2 ANC: skin (Infections and infestations) | 2
Hyperkalemia (Investigations) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Neurop: hear & bal. (Nervous system disorders) | 1
Hyponatremia (Investigations) | 10
Hyperuricemia (Investigations) | 3
Edema-trunk/genital (Blood and lymphatic system disorders) | 1
Musculo. Pain: joint (Musculoskeletal and connective tissue disorders) | 2
Lung Pain: chest/thorax (Respiratory, thoracic and mediastinal disorders) | 1
Musculo. Pain: limb (Musculoskeletal and connective tissue disorders) | 4
Edema-Head and Neck (Blood and lymphatic system disorders) | 1
Eye Infection Unk ANC: conjuct. (Eye disorders) | 1
Lung Pain: throat/phar/lar (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (Nervous system disorders) | 5
Hypotension (Cardiac disorders) | 4
Insomnia (General disorders) | 5
Mucositis, clin: oral cavity (Gastrointestinal disorders) | 6
Airway obstruction: trachea (Respiratory, thoracic and mediastinal disorders) | 1
Watery eye (Eye disorders) | 2
Bicarbonate, serum low (Investigations) | 2
Rhinitis (Immune system disorders) | 4
Hemorrhoids (Gastrointestinal disorders) | 2
GI Pain: anus (Gastrointestinal disorders) | 1
Memory impairment (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Tremor (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 4
Blood-other (Blood and lymphatic system disorders) | 3
Neuro Pain: neuralg/periph nrv (Nervous system disorders) | 1
Anorexia (Gastrointestinal disorders) | 7
Hypomagnesemia (Investigations) | 3
Eye inf, 0-2 ANC: conjunct. (Eye disorders) | 1
Dehydration (Gastrointestinal disorders) | 4
GI Pain: abdomen (Gastrointestinal disorders) | 3
Diplopia (Eye disorders) | 1
GI Inf, 0-2 ANC: stomach (Gastrointestinal disorders) | 1
Nasal/Paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Musculo. Pain: back (Musculoskeletal and connective tissue disorders) | 2
Bilirubin (Investigations) | 1
Muscle weakness: whole body (Musculoskeletal and connective tissue disorders) | 1
Liver dysfunction (Hepatobiliary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Skin Inf, 0-2 ANC: lip/perior (Infections and infestations) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Supra Arrhyth: supra tachy (Cardiac disorders) | 1
GI-other (Gastrointestinal disorders) | 1
Musculo. Pain: muscle (Musculoskeletal and connective tissue disorders) | 6
Creatinine (Investigations) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Hypernatremia (Investigations) | 3
Metabolic/Lab-other (Investigations) | 4
PTT (Investigations) | 2
Coagulation-other (Investigations) | 2
Musculo Pain: neck (Musculoskeletal and connective tissue disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Dermatology-other (Skin and subcutaneous tissue disorders) | 2
Salivary gland changes (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Acute vascular leak syndrome (Vascular disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 20
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Lung Pain: chest wall (Respiratory, thoracic and mediastinal disorders) | 2
cTnI (Investigations) | 1
Cardiac-general-other (Cardiac disorders) | 2
INR (Investigations) | 1
Acidosis (Investigations) | 1
Hypoglycemia (Investigations) | 1
Mucositis, clin: esophagus (Gastrointestinal disorders) | 2
Mood alteration: anxiety (Nervous system disorders) | 3
GI Inf, 0-2 ANC: gums (Infections and infestations) | 1
CPK (Investigations) | 1
Muscle weakness: low extrem (Musculoskeletal and connective tissue disorders) | 1
Cholesterol (Investigations) | 1
Gait/Walking (Musculoskeletal and connective tissue disorders) | 2
GI hemorrhage: lower GI (Gastrointestinal disorders) | 1
GI Inf, 0-2 ANC: abdomen NOS (Gastrointestinal disorders) | 1
GGT (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other